CLINICAL TRIAL: NCT00208416
Title: Randomised, Prospective, Post-Market Surveillance Study Comparing the Outcomes of Minimally Invasive and Conventional Surgical Procedures in Subjects Requiring Primary Total Hip Arthroplasty for Osteoarthritis.
Brief Title: A Randomised Multi-centre Study to Compare the Short-term Outcomes of Minimally Invasive and Conventional Surgery in Primary Total Hip Replacement
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Combination of departure of Investigator from one site and slow recruitment rate
Sponsor: DePuy International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CT02/29
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-03

CONDITIONS: Osteoarthritis(Primary)
Keywords: Hip; Surgical Technique

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): DePuy MI System
  Interventions: Procedure: DePuy MI System
- 2 (Active Comparator): Conventional surgical technique
  Interventions: Procedure: Conventional surgical technique

INTERVENTIONS:
Procedure: DePuy MI System — A minimally invasive surgical technique used in total hip replacement.
  Arms: 1
Procedure: Conventional surgical technique — A conventional surgical technique used in total hip replacement
  Arms: 2

SUMMARY:
The purpose of this study is to compare the short-term outcomes of two surgical techniques, minimally invasive and conventional, when used in the treatment of patients with hip joint disease requiring a total hip replacement. Patients who enter the study will be randomly allocated to undergo surgery using the minimally invasive or conventional surgical technique and will be evaluated at regular intervals following hip surgery using patient, clinical and x-ray assessments with a focus on short term rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

i) Male or female subjects, aged between 18 and 75 years inclusive.

ii) Subjects who are able to give voluntary, written informed consent to participate in this investigation and from whom consent has been obtained.

iii) Subjects who in the opinion of the Investigator, are able to understand this investigation, co-operate with the investigational procedures and are willing to return to the hospital for all the required post-operative follow-ups.

iv) Subjects with a primary diagnosis of osteoarthritis.

v) Subjects considered suitable for a primary total hip arthroplasty and are considered suitable for a minimally invasive surgical procedure.

Exclusion Criteria:

i) Subjects who, in the opinion of the Investigator, have an existing condition that would compromise their participation and follow-up in this study, or extend their time to discharge beyond that required for their hip replacement surgery.

ii) Women who are pregnant.

iii) Subjects who are known drug or alcohol abusers or with psychological disorders that could effect follow-up care or treatment outcomes.

iv) Subjects who have participated in a clinical study with an investigational product in the last 6 month(s).

v) Subjects who are currently involved in any injury litigation claims.

vi) Subjects with a Body Mass Index (BMI) > 30.

vii) Subjects with a malunion, arthrodesis or severe dysplasia with superior femoral head migration.

viii) Subjects requiring a simultaneous bilateral total hip arthroplasty.

ix) Subjects undergoing the second stage of a staged bilateral who are less than 9 months post-arthroplasty

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2005-10; Primary Completion 2007-12 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Number of hours post-operatively after which subjects are first able to mobilise with a frame or crutches | First post-operative day
Level of assistance required to perform 3 functional tasks (supine to sit, sit to stand and bed to chair transfer)on the second post-operative day | Second post-operative day
Time taken (in seconds) for subjects to walk 10 metres on the second post-operative day. | Second post-operative day
Amount of time (in seconds) for which subjects are able to stand on the operative leg on the second post-operative day. | Second post-operative day

SECONDARY OUTCOMES:
Haematological parameters assessed over a 56 hours post op | 56 hours post-operatively
Pain levels and wound condition | Until discharge
Trendelenberg sign | Until discharge and at 6 weeks
Day of discharge | Until discharge
Activity levels over specified distances | Until discharge
Harris Hip score | 6 weeks, 6 months, 1 yr, 2 yrs, 5 yrs and 10 yrs post-surgery
Oxford Hip score | 6 weeks, 6 months, 1 yr, 2 yrs, 5 yrs and 10 yrs post-surgery
Radiological analysis | 6weeks, 6mths, 1yr, 2yrs, 5yrs and 10yrs post-surgery

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Rotherham General Hospitals NHS Trust, Rotherham, South Yorkshire
  - Warwick Hospital NHS Trust, Warwick